CLINICAL TRIAL: NCT01888484
Title: Clinical Phase III Study to Evaluate the Pharmacokinetics, Efficacy, Tolerability and Safety of Subcutaneous Human Immunoglobulin (Octanorm 16.5%) In Patients With Primary Immunodeficiency Diseases
Brief Title: Study of Octanorm Subcutaneous IG in Patients With PID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCGAM-01
Record Dates: First submitted 2013-06-21; First posted 2013-06-27 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octanorm 16.5% (Experimental): octanorm 16.5%, human normal immunoglobulin for subcutaneous (SC) administration.
  Interventions: Biological: octanorm 16.5%

INTERVENTIONS:
Biological: octanorm 16.5% — octanorm 16.5%, human normal immunoglobulin for subcutaneous (SC) administration.

SUMMARY:
This is an open-label phase III study with a 12-week wash-in/wash-out period followed by a 12-month efficacy period. The main goals of the study are to assess the efficacy of octanorm in preventing serious bacterial infections (SBI) compared with historical control data and to evaluate the pharmacokinetic (PK) characteristics of octanorm.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 2 years up to and including 75 years.
2. Confirmed diagnosis of PI as defined by the ESID and PAGID and requiring immunoglobulin replacement therapy due to hypogammaglobulinaemia or agammaglobulinaemia. The exact type of PI should be recorded.
3. Patients with at least 6 infusions on regular treatment with any IVIG, there of a minimum of the last 2 months on the same product prior to entering the study. Constant IVIG dose between 200 and 800 mg/kg body weight (±20% of the mean dose for the last 6 infusions).
4. Availability of the IgG trough levels of 2 previous IVIG infusions before enrollment, and maintenance of greater than or equal to 5.0 g/L in the trough levels of these 2 previous infusions.
5. Negative result on a pregnancy test (HCG-based assay in urine) for women of childbearing potential and use of a reliable method of contraception for the duration of the study.
6. For adult patients: freely given written informed consent. For minor patients: freely given written informed consent from parents/legal guardians and written informed assent from the child/adolescent in accordance with the applicable regulatory requirements.
7. Willingness to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

Exclusion Criteria:

1. Acute infection requiring intravenous antibiotic treatment within 2 weeks prior to and during the screening period.
2. Known history of adverse reactions to IgA in other products.
3. Patients with body mass index ≥40 kg/m2.
4. Exposure to blood or any blood product or plasma derivatives, other than IVIG treatment for PID, within the past 3 months prior to the first infusion of octanorm.
5. Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products, or any component of the investigational product (such as Polysorbate 80).
6. Requirement of any routine premedication for IgG administration.
7. History of malignancies of lymphoid cells and immunodeficiency with lymphoma.
8. Severe liver function impairment (ALAT 3 times above upper limit of normal).
9. Known protein-losing enteropathies or proteinuria.
10. Presence of renal function impairment (creatinine greater than 120 uM/L), or creatinine greater than 1.35 mg/dL), or predisposition for acute renal failure (e.g., any degree of pre-existing renal insufficiency or routine treatment with known nephritic drugs).
11. Treatment with oral or parenteral steroids for greater than or equal to 30 days or when given intermittently or as bolus at daily doses greater than or equal to 0.15 mg/kg.
12. Treatment with immunosuppressive or immunomodulatory drugs.
13. Live viral vaccination (such as measles, rubella, mumps and varicella) within the last 2 months prior to first infusion of octanorm.
14. Treatment with any investigational medicinal product within 3 months prior to first infusion of octanorm.
15. Presence of any condition, that is likely to interfere with the evaluation of study medication or satisfactory conduct of the trial.
16. Known or suspected to abuse alcohol, drugs, psychotropic agents or other chemicals within the past 12 months prior to first infusion of octanorm.
17. Known or suspected HIV, HCV, or HBV infection.
18. Pregnant or nursing women.
19. Planned pregnancy during the course of the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-03; Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Study Director — International Medical Director
Locations (23):
- United States (7):
  - Octapharma Research Site, Birmingham, Alabama
  - Octapharma Research Site, Irvine, California
  - Octapharma Research Site, San Diego, California
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, Omaha, Nebraska
  - Octapharma Research Site, Toledo, Ohio
  - Octapharma Research Site, Frisco, Texas
- Canada (2):
  - Octapharma Research Site, Edmonton
  - Octapharma Research Site, Montreal
- Czechia (4):
  - Octapharma Research Site, Brno
  - Octapharma Research Site, Olomouc
  - Octapharma Research Site, Pilsen
  - Octapharma Research Site, Prague
- Octapharma Research Site, Budapest, Hungary
- Poland (3):
  - Octapharma Research Site, Bialystok
  - Octapharma Research Site, Krakow
  - Octapharma Research Site, Lublin
- Russia (3):
  - Octapharma Research Site, Moscow
  - Octapharma Research Site, Saint Petersburg
  - Octapharma Research Site, Yekaterinburg
- Slovakia (3):
  - Octapharma Research Site, Bratislava
  - Octapharma Research Site, Košice
  - Octapharma Research Site, Martin

REFERENCES:
- [Derived] Kobayashi RH, Gupta S, Melamed I, Mandujano JF, Kobayashi AL, Ritchie B, Geng B, Atkinson TP, Rehman S, Turpel-Kantor E, Litzman J. Clinical Efficacy, Safety and Tolerability of a New Subcutaneous Immunoglobulin 16.5% (Octanorm [Cutaquig(R)]) in the Treatment of Patients With Primary Immunodeficiencies. Front Immunol. 2019 Feb 4;10:40. doi: 10.3389/fimmu.2019.00040. eCollection 2019. PMID 30778345

RESULTS

PARTICIPANT FLOW:
Groups:
- Children ≥2 Years <6 Years: Children ≥2 Years <6 Years
- Children Aged ≥6 to <12 Years: Children Aged ≥6 to <12 years
- Adolescents ≥12 Years <17 Years: Adolescents ≥12 Years <17 Years
- Adults ≥17 Years ≤75 Years: Adults ≥17 Years ≤75 Years
Period: Overall Study
Arm/Group | Children ≥2 Years <6 Years | Children Aged ≥6 to <12 Years | Adolescents ≥12 Years <17 Years | Adults ≥17 Years ≤75 Years
Started | 12 | 14 | 12 | 37
Completed | 12 | 14 | 8 | 34
Not Completed | 0 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients.
  The data are reported as the overall population as it was not the intent of the protocol to report analysis by age group
Arm/Group | All Patients
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.81 (21.911)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 74
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of SBI Per Person-year
Description: The primary efficacy outcome is the rate of SBI (Serious bacterial infections - defined as bacteremia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, and visceral abscess) per person-year on treatment.
Time Frame: Every 4 weeks until the final evaluation at week 65.
Population: The data are reported as the overall population as it was not the intent of the protocol to report analysis by age group
Measure: Number; unit: SBIs per person year
Groups:
- All Patients: All patients
Arm/Group | All Patients
Number analyzed (Participants) | 75
SBIs per person year | 0

2. Primary Outcome: AUC(t) at Steady-State Conditions
Description: The primary endpoint with respect to the PK investigations is the area under the curve AUC(t) (i.e., AUC from time 0 (start of the infusion) to the end of the nominal dosing period, standardised to 1 week) at PKSC2 at steady-state conditions.
Time Frame: Measured at Week 28 before the start of the SC infusion, 10 minutes before the end of the infusion, and at 2 h, 1, 2, 3, 4 and 7 days after the end of the infusion. Calculated and averaged.
Population: In several cases, AUCτ could not be calculated due to very flat time-concentration profiles.
Measure: Mean (Standard Deviation); unit: h*g/L
Groups:
- Total Patients: All patients
Arm/Group | Total Patients
Number analyzed (Participants) | 24
h*g/L | 2232.61 (585.842)

3. Secondary Outcome: The Annual Rate of All Infections of Any Kind or Seriousness.
Description: The annual rate of all infections of any kind or seriousness.
Time Frame: Up to 65 weeks
Population: as for outcome 1
Measure: Number; unit: infections per person-year
Arm/Group | Total Patients
Number analyzed (Participants) | 75
infections per person-year | 3.414

4. Secondary Outcome: Non-serious Infections
Description: Non-serious infections (total and by category).
Time Frame: Up to 65 weeks
Population: as for outcome 1
Measure: Number; unit: infections
Arm/Group | Total Patients
Number analyzed (Participants) | 75
infections
  Ear infections | 8
  Eye infections | 3
  Infections of the GI tract | 25
  Infections of the genitourinary tract | 24
  Upper respiratory tract infections | 179
  Lower respiratory tract infections | 32
  Infections of the skin | 6
  Infections not (elsewhere) classified | 16

5. Secondary Outcome: Cmax of Total IgG and IgG Subclasses
Description: Cmax (Maximum Plasma Concentration) of total IgG and IgG Subclasses, where the mean value was calculated and reported
Time Frame: Measured at week 28
Population: The data are reported as the overall population as it was not the intent of the protocol to report analysis by age group. Data not available for all patients.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | All Patients
Number analyzed (Participants) | 37
g/L
  IgG Total Cmax | 13.47 (3.655)
  IgG1 Cmax | 8.56 (1.858)
  IgG2 Cmax | 3.88 (1.532)
  IgG3 Cmax | 0.32 (0.127)
  IgG4 Cmax | 0.40 (0.567)

6. Secondary Outcome: Tmax of Total IgG and IgG Subclasses
Description: Tmax (Time to Maximum Plasma Concentration) of total IgG and IgG Subclasses
Time Frame: Measured at Week 28 for all patients, median value was calculated
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | All Patients
Number analyzed (Participants) | 37
hours
  Tmax Total IgG | 49.62 [0.8 to 98.3]
  Tmax IgG1 | 50.50 [1.5 to 167.7]
  Tmax IgG2 | 72.20 [0.5 to 167.7]
  Tmax IgG3 | 49.62 [1.8 to 98.1]
  Tmax IgG4 | 47.50 [0.6 to 167.7]

7. Secondary Outcome: AUC of Total IgG and IgG Subclasses
Description: AUC (Area Under the Concentration-Time Curve) of total IgG and IgG Subclasses calculated for all patients and mean value was calculated and reported
Time Frame: Measured at Week 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*g/L
Arm/Group | All Patients
Number analyzed (Participants) | 25
hr*g/L
  IgG Total AUC: number analyzed (Participants) | 24
  IgG Total AUC | 2232.61 (585.842)
  IgG1 AUC: number analyzed (Participants) | 22
  IgG1 AUC | 1424.69 (298.776)
  IgG2 AUC: number analyzed (Participants) | 23
  IgG2 AUC | 659.57 (262.295)
  IgG3 AUC | 48.65 (18.455)
  IgG4 AUC | 71.40 (102.578)

8. Secondary Outcome: Trough Levels of Serum IgG
Description: Trough levels of serum IgG, IgG1, IgG2, IgG3, IgG4 at PK 7 days after 28th infusion of octanorm measured for all patients and median value was calculated and reported
Time Frame: Measured once at Week 28, seven days after 28th infusion of octanorm
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | All Patients
Number analyzed (Participants) | 36
g/L
  Total IgG | 11.85 [10.00 to 13.70]
  IgG1 | 7.51 [6.58 to 9.00]
  IgG2 | 3.12 [2.69 to 3.85]
  IgG3 | 0.27 [0.20 to 0.34]
  IgG4 | 0.15 [0.11 to 0.32]

9. Secondary Outcome: IVIG to Octanorm DCF (Based on the Area Under the Concentration-time Curve [AUCτ])
Description: IVIG to Octanorm Dose Conversion Factor (based on the area under the concentration-time curve [AUCτ]) -- determined by least-squares regression Model which was without restriction of the intercept.
Time Frame: AUC Measured at Week 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | All Patients
Number analyzed (Participants) | 37
unitless | 1.278 (0.9401)

ADVERSE EVENTS:
Time Frame: For the duration of the 65 week treatment period starting with the first infusion of octanorm.
Description: The data are reported as the overall population as it was not the intent of the protocol to report analysis by age group
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 9/75
Other Adverse Events (participants affected / at risk) | 61/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=75)
Abscess limb (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Acute odontogenic jaw osteomyelitis (Infections and infestations) | 1 (1)
Pneumocystitis jiroveci infection (Infections and infestations) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asperger's syndrome (Psychiatric disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=75)
Leukopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Headache (Nervous system disorders) | 6 (14)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Diarrhoea (Gastrointestinal disorders) | 11 (18)
Vomiting (Gastrointestinal disorders) | 6 (8)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Pyrexia (General disorders) | 12 (14)
Arthropod bite (Injury, poisoning and procedural complications) | 8 (9)
Excoriation (Injury, poisoning and procedural complications) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Acute sinusitis (Infections and infestations) | 5 (13)
Bronchitis (Infections and infestations) | 7 (14)
Gastroenteritis viral (Infections and infestations) | 4 (6)
Influenza (Infections and infestations) | 5 (5)
Laryngitis (Infections and infestations) | 4 (5)
Nasopharyngitis (Infections and infestations) | 17 (37)
Otitis media (Infections and infestations) | 4 (5)
Rhinitis (Infections and infestations) | 11 (17)
Rhinovirus infection (Infections and infestations) | 5 (7)
Sinusitis (Infections and infestations) | 15 (25)
Upper respiratory tract infection (Infections and infestations) | 21 (33)
Urinary tract infection (Infections and infestations) | 6 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dysuria (Renal and urinary disorders) | 4 (4)
Any infusion site reaction (Skin and subcutaneous tissue disorders) | 55 (994)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT01888484/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT01888484/SAP_001.pdf